CLINICAL TRIAL: NCT07002372
Title: Impact of Procedural Video Viewing on Patients Undergoing Intravitreal Anti-VEGF Injections
Brief Title: Effect of Video Viewing on Intravitreal Injection Experience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-1393
Record Dates: First submitted 2025-05-20; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Age Related Macular Degeneration; Diabetic Retinopathy; Choroidal Neovascularization; Retinal Vein Occlusion; Cystoid Macular Edema
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Choroidal Neovascularization; Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procedural video viewing Group (Experimental): Participants will watch an educational video explaining the injection procedure prior to treatment.
  Interventions: Behavioral: Procedure video viewing
- Control Group (No Intervention): Participants will not view the video before the treatment.

INTERVENTIONS:
Behavioral: Procedure video viewing — Patients who have never had an intravitreal injection before will be randomly assigned to watch an educational video about the procedure prior to treatment.
  Arms: Procedural video viewing Group

SUMMARY:
Study Objective The goal of this clinical trial is to evaluate whether viewing a procedural video can improve the patient experience and reduce the incidence and severity of subconjunctival hemorrhage in individuals undergoing intravitreal anti-VEGF injections.

Key Research Questions

1. Can viewing the procedural video prior to treatment reduce the rate and/or area of subconjunctival hemorrhage?
2. Can the video improve the patient experience, specifically by reducing anxiety levels and increasing satisfaction with the treatment process?

Study Design Participants will be randomly assigned to either an intervention group, who will watch an educational video explaining the injection procedure, or a control group, who will not view the video.

All participants will complete the State-Trait Anxiety Inventory-State (STAI-S) questionnaire both before and after treatment to assess changes in anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving their first intravitreal injection of anti-VEGF medication due to retinal diseases
* Mentally competent, and able to communicate without barriers
* Willing to voluntarily sign an informed consent form.

Exclusion Criteria:

* History of previous eye surgery
* Best-corrected visual acuity in the better eye worse than 0.3
* The target eye is complicated with neovascular glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Rate and area of subconjunctival hemorrhage | 3 minutes after the intravitreal injection procedure.
  After the injection, a photograph of the eye will be taken to document the presence of subconjunctival hemorrhage and to measure the hemorrhage area using ImageJ software.

SECONDARY OUTCOMES:
Anxiety levels assessed by State-Trait Anxiety Inventory-State (STAI-S) | 30 minutes before and after the procedure.
  State-Trait Anxiety Inventory-State (STAI-S) questionnaire both before and after treatment to assess changes in anxiety levels

OTHER OUTCOMES:
Patient satisfaction assessed by a satisfaction score questionnaire | 30 minutes after the procedure.
  Patient satisfaction with the treatment process will be assessed using a 10-point Likert scale satisfaction score collected after the procedure, where 1 indicates "not satisfied at all" and 10 indicates "completely satisfied".
Physician's assessment of patient cooperation during the procedure | Immediately after the intravitreal injection procedure
  Physician's assessment of patient cooperation during the procedure Patient cooperation will be assessed by the physician immediately after the procedure using a 10-point Likert scale, where 1 indicates completely uncooperative and 10 indicates fully cooperative. The scale is based on observable patient behavior such as adherence to instructions, physical movements, and verbal interaction during the procedure.
Total procedure time | During the procedure.
  The time duration from the start of disinfection to the completion of the injection.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Fang, MD., PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Yahalomi T, Hecht I, Lagstein O, Nemet A, Pe'er L, Hadad F, Keren-Yaar A, Kassem R, Burgansky-Eliash Z, Bar A, Achiron A. REDUCTION OF POSTINTRAVITREAL INJECTION PAIN USING ICE: An Open-Label Interventional Randomized Controlled Trial. Retina. 2020 Jul;40(7):1434-1438. doi: 10.1097/IAE.0000000000002608. PMID 31305506
- [Background] Boyle J, Vukicevic M, Koklanis K, Itsiopoulos C, Rees G. Experiences of patients undergoing repeated intravitreal anti-vascular endothelial growth factor injections for neovascular age-related macular degeneration. Psychol Health Med. 2018 Feb;23(2):127-140. doi: 10.1080/13548506.2016.1274040. Epub 2017 Jan 9. PMID 28064517